CLINICAL TRIAL: NCT07143851
Title: Research on Key Technologies of Intelligent Auxiliary Diagnosis for Multiple Eye Diseases Based on Multimodal Ultra-High-Speed SS-OCT/OCTA
Brief Title: Multi-modal Intelligent Diagnosis System for Multiple Ophthalmic Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BJ-2025-092
Record Dates: First submitted 2025-07-29; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Retina Disease; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

INTERVENTIONS:
Other: Not applicable- observational study — There is no special intervention method

SUMMARY:
Aiming at the problems of low image reading efficiency, crowded medical resources and fragmented cross-modal information of ophthalmic OCT and OCTA, a multimodal large model diagnostic framework for various diseases such as retinal diseases and optic nerve damage in glaucoma is constructed to fully explore the complementary information of various images such as SS-OCT structural images, SS-OCTA vascular images and optic nerve scans. Extract cross-modal joint features to improve the accuracy of automatic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as macular degeneration, diabetic macular edema, retinal vein obstructive macular edema, high myopia, glaucoma or other clearly diagnosed ophthalmic diseases. The SS-OCT/SS-OCTA images of the patient are clear.

Exclusion Criteria:

* The image quality is poor and difficult to analyze due to reasons such as refractive media opacity and poor coordination.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as macular degeneration, diabetic macular edema, retinal vein obstructive macular edema, high myopia, glaucoma or other clearly diagnosed ophthalmic diseases.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
CMT | Baseline
  Central macular thickness measured on OCT

SECONDARY OUTCOMES:
SS-OCT/OCTA images | Baseline
  Multimodal features based on patients' iamges

IPD SHARING:
Plan to Share IPD: No